CLINICAL TRIAL: NCT01716442
Title: A Multi-center Randomized Controlled Trial of Rituximab for Refractory Nephrotic Syndrome in Children
Brief Title: Rituximab Trial for Pediatric Nephrotic Syndrome
Acronym: RTX2012
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Childrens Hospital (Other)
Responsible Party: Principal Investigator, Hee Gyung Kang, Associate Professor, Seoul National University Childrens Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTX-2012
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Steroid Resistant Nephrotic Syndrome; Steroid Dependent Nephrotic Syndrome
Keywords: rituximab; nephrotic; refractory
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- steroid-resistant (Active Comparator): Steroid-resistant group: n=27 , enroll all for treatment
  Interventions: Drug: Rituximab
- steroid-dependent-rituximab (Active Comparator): steroid-responsive group: n=38
  Interventions: Drug: Rituximab
- steroid-dependent-placebo (Placebo Comparator): steroid-responsive group: n=23
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Per dose: Rituximab 375 mg/m2 (max.500mg/day). efficacy monitored by CD19 cell count. If CD19 cells are not depleted, second or third doses are given at 2-3 weeks interval.
  Other Names: Mabthera; 2005110300291 (rituximab)
  Arms: steroid-dependent-rituximab; steroid-resistant
Drug: Placebo
  Arms: steroid-dependent-placebo

SUMMARY:
Anti-CD20 agent has been proposed as a rescue therapy for refractory nephrotic syndrome(NS) on the basis of favorable clinical observations. Yet the long-term effect on maintaining remission or the likelihood of becoming rituximab-dependent is unclear and the information on the safety profile of rituximab is limited. This trial was designed to investigate the safety and efficacy of Rituximab in children with refractory NS.

ELIGIBILITY:
Inclusion Criteria:

(A)steroid/calcineurin inhibitor resistant nephrotic syndrome

1. steroid resistance: no remission after 4 weeks of daily oral corticosteroid (60mg/m2/day)
2. calcineurin inhibitor resistance: no remission after 3 months of therapeutic dose administration of cyclosporine and/or tacrolimus
3. no remission defined by persistent proteinuria of nephrotic range for the last 3 months
4. post-transplant patients were included in the study

(B)steroid-dependent nephrotic syndrome

1. Steroid-dependent patients who had been on various known medications (such as corticosteroids, cyclophosphamide, chlorambucil, calcineurin inhibitors, levamisole ..) continuously for more than 2 years
2. definition of dependency: more than two consecutive relapse events in 2 weeks after discontinuation of steroid or calcineurin inhibitor

   * no improvement in relapsing frequency with calcineurin inhibitor use
   * unable to continue with calcineurin inhibitor due to side effects
   * unable to continue with calcineurin inhibitor due to prolonged use (over 2 years)
   * other conditions in which the clinician considers difficult to control disease with steroids or calcineurin inhibitors only.

Exclusion Criteria:

* previous rituximab use
* secondary nephrotic syndrome
* estimated GFR <60mL/min/1.73m2 or under 50% of age-matched standard GFR
* chronic or acute active infection (e.g. hepatitis B,C, herpes, varicella zoster)
* prior live vaccine inoculation within 1 month (from the study enrollment)
* cardiovascular diseases, pulmonary or pleural diseases
* uncontrolled hypertension
* leukocytopenia (absolute neutrophil count <1500/mm3) or thrombocytopenia (<75000/mm3)
* pregnancy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
The remission rate of steroid-resistant nephrotic syndrome patients after rituximab treatment | within 6 months from the initiation of treatment
The rate of maintaining remission in steroid-dependent nephrotic syndrome patients | within 6 months from the initiation of treatment versus placebo control

CONTACTS AND LOCATIONS:
Overall Officials: Hee Gyung Kang A. Kang, M.D., Ph.D., Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526